CLINICAL TRIAL: NCT07202351
Title: Impact of an Intervention Targeting Sleep Disorders During Tobacco or Cannabis Cessation Therapy: a Randomised Pilot Study
Brief Title: Targeted Intervention on Sleep Disorders During Tobacco or Cannabis Cessation Therapy
Acronym: ISAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Principal Investigator, Pierre Alexis GEOFFROY, University professor and Hospital practitioner, Centre Hospitalier St Anne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D22_EPI0029
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disorder
Keywords: sleep disorder; tobacco; cannabis; addiction
MeSH Terms: conditions — Sleep Wake Disorders; Marijuana Abuse; Behavior, Addictive | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: Randomised pilot clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contrôle (No Intervention): In the control group, patients benefit from care as usual in one of the two addiction prevention and care clinics.
- Intervention (Experimental): In the intervention group, patients will be benefit, in addition to the usual care of the smoking / tobacco cessation therapy, from a specific intervention to screen and care for sleep disorders, at the Chronos centre.
  Interventions: Other: Screening and management of sleep disorders

INTERVENTIONS:
Other: Screening and management of sleep disorders — Patients in the intervention group will undergo a systematic and standardised screening of sleep disorders. If any trouble is identified, a specific treatment plan is offered at the Chronos centre, including for instance, cognitive behavioural therapy for insomnia, or nightmares will be treated with Image Rehearsal Therapy (IRT).
  Arms: Intervention

SUMMARY:
During a cessation therapy for tobacco or cannabis, sleep disorders are one of the main risk factors of relapse, and a symptom of substance withdrawing. In this study, we make the hypothesis that identifying and managing potential sleep disorders during cessation treatment may contribute to maintain tobacco / cannabis abstinence on the long-term. To evaluate the impact of such intervention, we will conduct a randomised pilot study among patients consulting at two addiction prevention and care centres, for smoking or cannabis use cessation treatment. Control group will benefit of usual care (a multidisciplinary care with individual and group therapies); intervention group will benefit in addition of a systematic screening of sleep disorders, and in case of a diagnosed alteration, they will be addressed to the Chronos centre, for specific care to help them manage and reduce the consequences of their sleep disorders. Participants will be followed over a 6-month period, with visits at 1 and 3 months, to monitor smoking or cannabis cessation, and other criteria associated with their substance use or sleep.

DETAILED DESCRIPTION:
Smoking is a serious public health issue in France, with one quarter of the population who smokes on a daily base. Tobacco use represents the first avoidable death cause. Cannabis, often use with tobacco, is the most frequent drug use, worldwide and with a prevalence of 3.2% of regular users in France, including 2.1% of daily users. Both substances are associated with sleep disorders; for instance, nicotine has several side effects, such as a negative impact on sleep quality and structure. During cessation therapy, sleep disorders were identified as a risk factor of relapse and one of the main lasting symptoms. Therefore, relation between addiction and sleep disorders seem to be bidirectional, potentially increasing the impact of each other. Screening and managing sleep disorders as a preventive measure to avoid relapse represents an improvement during smoking or cannabis use cessation treatment.

The main objective of the study is to evaluate the impact of a specific intervention targeting sleep disorders during tobacco or cannabis cessation therapy. We will conduct a randomised pilot study among patients presenting at two participating addiction prevention and care centres, for smoking or cannabis use cessation treatment. Patients who are eligible and agree to participate will be randomised in either control group, and will benefit of the usual care, or intervention group, and will benefit in addition of a systematic and standardised screening of sleep disorders, and specific care at the Chronos centre, if any disorder is diagnosed.

Patients will be followed over a 6-month period, with two visits at 1 and 3 months, to monitor indicators related to substance consumption and sleep. The impact of the targeted intervention will be evaluate based on the abstinence duration over the 6 months, calculated on the total number of days without tobacco / cannabis use. We will also collect other information that can be associated with the success or failure of cessation therapy, such as depressive symptoms, anxiety disorders, the use of other psychoactive substances (alcohol for instance), other psychiatric disorder, etc.

Questions on sleep will be asked to patients in the control group, to assess comparability of both groups throughout the study. This pilot trial will allow us to determine the feasibility and efficacy of a targeted intervention on sleep disorders during smoking or cannabis use cessation therapy, in order to generalise such care in the usual practice.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* presenting at the participating addiction treatment centres for a smoking or cabannis use cessation therapy
* who agree to participate to the study
* affiliated to the French health insurance system

Exclusion Criteria:

* Patients hospitalised during the cessation therapy
* Patients undergoing sleep disorders treatment
* Patients participating to another study
* Patients with psychotic disorders (according the DSM-5 classification)
* Patients who do not want the additionnal intervention and care if randomised in the intervention group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Abstinence | M6: 6 months after inclusion
  Abstinence to the substance (tobacco or cannabis, or both) defined by the absence of use of tobacco / cannabis products over the 6 month period after inclusion. Abstinence will be assessed with the Timeline Followback (TLFB), a self-reported calendar of substance consumption.

SECONDARY OUTCOMES:
Relapse | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Relapse rate. Relapse is defined as ≥ 7 consecutive days of smoking tobacco or cannabis. Relapse will be assessed with the Timeline Followback (TLFB), a self-reported calendar of substance consumption.
Abstinence number of days | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Longest period (number of consecutive days) without substance use, which will be assessed with the Timeline Followback (TLFB), a self-reported calendar of substance consumption.
Consumption number of days | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Longest period (number of consecutive days) with substance use, which will be assessed with the Timeline Followback (TLFB), a self-reported calendar of substance consumption.
Carbon monoxide | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Exhaled carbon monoxide test to monitor CO to assess objectively smoking level
Insomnia | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  The severity of insomnia will be measured with the Insomnia Severity Index (ISI). Total score ranges from 0-28. INterpretation of the score 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Sleep quality | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). Total score ranges form 0 (better) to 21 (worse) sleeping quality.
Sleepiness | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Sleepiness will be evaluated with the Epworth Sleepiness Scale, which ranges from 0 to 24. Results from 0 to 10 show average (normal) daytime sleepiness and from 11 to 24 indicates excessive (abnormal) daytime sleepiness.
Medication | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Patients will be asked if they take any medication to help reduce their sleep disorders (hypnotics, melatonin, etc.).
Anxiety and depression | M1: 1 month after inclusion M3: 3 months after inclusion M6 : 6 months after inclusion
  Anxiety and depressive symptoms will be assessed using the Hospital Anxiety and Depression scale (HADs).
  There are two scores for items in each subscale : anxiety score (HADS-A) and depression score (HADS-D). Total score ranging from 0-21 for each subscale. A higher score indicates higher distress. Usually, a cut-off score of 11 for the total HADS, and 8 for the HADS-D are used.

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris Psychiatrie et Neurosciences, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided upon reasonable request addressed to the investigators.